CLINICAL TRIAL: NCT00098917
Title: A Phase I Clinical Trial of Mature Autologous Dendritic Cells Loaded With Irradiated Autologous Tumor Cells for the Treatment of Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Vaccine Therapy in Treating Patients Who Are Undergoing Surgery for Stage IB, Stage II, or Stage IIIA Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000396774; UCLA-0406031-01; NCI-6766
Record Dates: First submitted 2004-12-08; First posted 2004-12-09 (Estimated); Last update posted 2008-01-28 (Estimated); Status verified 2007-04

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — FANG vaccine; Chemotherapy, Adjuvant; Biological Therapy; Surgical Procedures, Operative; Immunotherapy, Active

INTERVENTIONS:
Drug: autologous tumor cell vaccine
Drug: therapeutic autologous dendritic cells
Procedure: adjuvant therapy
Procedure: biological therapy
Procedure: conventional surgery
Procedure: surgery
Procedure: tumor cell derivative vaccine
Procedure: vaccine therapy

SUMMARY:
RATIONALE: Vaccines made from a person's tumor cells and white blood cells may make the body build an effective immune response to kill tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of vaccine therapy in treating patients who are undergoing surgery for stage IB, stage II, or stage IIIA non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of adjuvant autologous dendritic cells loaded with irradiated autologous tumor cells in patients with stage IB-IIIA non-small cell lung cancer undergoing resection.
* Determine the safety and tolerability of this vaccine in these patients.

Secondary

* Determine the feasibility of this vaccine in these patients.
* Determine vaccine-specific and antitumor immunity in patients treated with this vaccine.

OUTLINE: This is a dose-escalation study.

Patients undergo leukaphersis to isolate peripheral blood mononuclear cells (PBMC). PBMC are expanded ex vivo to generate monocyte-derived dendritic cells (DC). Autologous tumor cells are harvested and purified at the time of surgical resection. DC are then loaded with irradiated autologous tumor cells.

Within 4-8 weeks after surgical resection, patients receive autologous DC loaded with irradiated autologous tumor cells intradermally on approximately days 1, 30, and 60 in the absence of unacceptable toxicity.

Cohorts of 6-9 patients receive escalating doses of vaccine until the maximum tolerated dose (MTD) is determined. If 2 of 9 patients in the first cohort experience dose-limiting toxicity, that dose level is considered the MTD.

Patients are followed at approximately 1 and 4 months, and then every 6 months for 4 years.

PROJECTED ACCRUAL: A total of 12-15 patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of non-small cell lung cancer

  * Clinical stage IB-IIIA disease
* Candidate for surgical resection as primary treatment for tumor

  * Surgically resectable tumor ≥ 2.0 cm in diameter
* No brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-1

Life expectancy

* Not specified

Hematopoietic

* Platelet count ≥ 100,000/mm^3
* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Hematocrit ≥ 30%

Hepatic

* Hepatitis B surface antigen negative*
* Hepatitis B core antigen negative*
* Hepatitis C virus negative*
* Bilirubin ≤ 2.0 mg/dL
* AST and ALT ≤ 2 times upper limit of normal NOTE: *Screening performed only if liver enzymes are elevated

Renal

* Creatinine ≤ 2.2 mg/dL
* BUN ≤ 40 mg/dL

Pulmonary

* FEV_1 > 2.0 L (pre-resection) OR
* Predicted post-resection FEV_1 > 1.0 L
* No more than 2 chronic obstructive pulmonary disease exacerbations requiring > 2 weeks of oral steroids and/or hospitalization within the past year

Immunologic

* Purified protein derivative (PPD) skin test negative
* HIV-1 and HIV-2 negative
* No acute infection, including any acute viral, bacterial, or fungal infection requiring specific therapy within the past 7 days
* No allergy to study agents
* No known autoimmune or collagen vascular disorder

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No underlying condition that would preclude study therapy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent anti-tumor necrosis factor agents

Chemotherapy

* Standard adjuvant chemotherapy for lung cancer allowed provided therapy is completed ≥ 30 days before administration of the first study vaccine
* No concurrent cyclophosphamide

Endocrine therapy

* No concurrent high-dose corticosteroids (e.g., > 10 mg of prednisone)
* Concurrent corticosteroids for minor breathing exacerbations allowed provided patient receives ≤ 2 short courses (≤ 10 days per course) within a 45-day period
* No concurrent corticosteroids within 48 hours before or after study vaccine administration

Radiotherapy

* Standard adjuvant radiotherapy for lung cancer allowed provided therapy is completed ≥ 30 days before administration of the first study vaccine

Surgery

* No prior organ allograft

Other

* No concurrent antihistamines within 48 hours before or after study vaccine administration
* No concurrent cimetidine or other H2 blockers within 48 hours before or after study vaccine administration
* Concurrent antibiotics for minor infection allowed provided patient receives ≤ 2 short courses (≤ 10 days per course) within a 45-day period
* No concurrent cyclosporine
* No concurrent azathioprine
* No other concurrent drugs known to significantly alter immune function
* No concurrent cytotoxic therapy
* No concurrent participation in another clinical trial involving experimental therapy
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2005-02

CONTACTS AND LOCATIONS:
Overall Officials: Michael D. Roth, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States